CLINICAL TRIAL: NCT06355024
Title: a Pilot Study to Explore the Efficacy of Inosine Reversing Chemo Resistance in Triple Negative Breast Cancer
Brief Title: Inosine Reverse Chemo Resistance in Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2024.1.30
Record Dates: First submitted 2024-03-30; First posted 2024-04-09 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Inosine; taxane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inosine (Experimental): oral inosine arm
  Interventions: Drug: Inosine; Drug: Taxane/Anthracycline/Eribulin Mesylate/Vinorelbine/Capecitabine/Carboplatin/UTD1/platinum

INTERVENTIONS:
Drug: Inosine — oral inosine 200mg tid
Drug: Taxane/Anthracycline/Eribulin Mesylate/Vinorelbine/Capecitabine/Carboplatin/UTD1/platinum — Taxane/Anthracycline/Eribulin Mesylate/Vinorelbine/Capecitabine/Carboplatin/UTD1/platinum

SUMMARY:
This is a Phase II, open-label, single-arm study evaluating the efficacy and safety of combined treatment of Inosine with chemotherapy in mTNBC (triple negative breast cancer) patients who progressed during previous chemotherapy.

DETAILED DESCRIPTION:
This is a Phase II, open-label, single-arm study evaluating the efficacy and safety of combined treatment of Inosine with chemotherapy in metastatic TNBC (triple negative breast cancer) patients who progressed during or following previous chemotherapy. Chemotherapy is the backbone drug for TNBC. How to reverse chemotherapy resistance or how to increase the sensitivity of chemotherapy efficacy, has become an urgent clinical problem to be solved. The preclinical results show that Inosine play a potentially important role in regulating the tumor microenvironment. The investigators found that inosine from intestinal probiotics was negatively correlated with breast cancer recurrence and metastasis after chemotherapy, and further functional experiments showed that inosine-producing flora or dietary supplementation with inosine could significantly inhibit the survival of tumor cells after chemotherapy and inhibit the recurrence and metastasis of breast cancer. Furthermore, it is considered to have a high level of safety. Based on preclinical studies, the investigators designed this study to enroll mTNBC patients who have progressed during or following chemotherapy, and to explore the efficacy of combined inosine with chemotherapy at a clinical level, providing new strategies of combined treatment for TNBC patients.

ELIGIBILITY:
Inclusion Criteria:

- ECOG Performance Status of 0, 1

* Metastatic or locally advanced, histologically documented TNBC (absence of HER2, ER, and PR expression)
* Radiologic/objective evidence of recurrence or disease progression after chemotherapy for metastatic breast cancer (MBC)
* Adequate hematologic and end-organ function, laboratory test results, obtained within 14 days prior to initiation of study treatment.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures as outlined for each specific treatment arm
* Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1)
* have the cognitive ability to understand the protocol and be willing to participate and to be followed up

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing CNS metastases
* Active or history of autoimmune disease or immune deficiency
* Significant cardiovascular disease
* History of malignancy other than breast cancer within 5 years prior to screening, with the exception of those with a negligible risk of metastasis or death
* Treatment with chemotherapy, radiotherapy,immunotherapy or surgery (outpatient clinic surgery excluded) within 3 weeks prior to initiation of study treatment.
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study
* History of allergies to the drug components of this trial
* Patients who have been using oral steroid hormones for a long time will need to stop for 4 weeks if they have used them occasionally in the past

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-05-11 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Baseline through end of study, assessed up to 6 months
Progression Free Survival (PFS) | Randomization to death from any cause, through the end of study,assessed up to 6 months
Biomarker analysis1 | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  The distribution of immune cells in pre- and post-treatment blood samples, alterations in gut microbiota in fecal samples, the infiltration of immune cells, and the proliferation and apoptosis of tumor cells in metastatic puncture samples.
Safety and treatment-related AEs | Randomization to death from any cause, through the end of study,assessed up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China